CLINICAL TRIAL: NCT05210569
Title: Visual Outcomes of the AcrySof® Vivity Intraocular Lens in Patients With High Ocular Axial Length
Brief Title: Visual Outcomes of Vivity in Patients With High Axial Length
Status: Completed | Type: Observational
Sponsor: Dr. James J. Wiens Medical Corporation (Other)
Collaborators: Sengi (Industry)
Responsible Party: Sponsor
Other Study IDs: JW-21-001
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Cataract
Keywords: EDOF IOL Vivity
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Bilateral implantation of the Vivity IOL: Vivity intraocular lens (IOL)
  Interventions: Device: Vivity

INTERVENTIONS:
Device: Vivity — Vivity intraocular lens (IOL)

SUMMARY:
The objective is to assess the visual outcomes and quality of vision of patients receiving the AcrySof® Vivity Intraocular lens (IOL), when implanted in eyes with high ocular axial length (≥24.5mm), after uneventful cataract surgery.

DETAILED DESCRIPTION:
This study is a single-arm unmasked clinical evaluation study of binocular uncorrected visual acuity at distance (6m), intermediate (66cm) and near (40cm), when implanted in eyes with high ocular axial length (≥24.5mm), after successful bilateral cataract surgery. Subjects will be assessed preoperatively, operatively, and at 1 day, 1 week, 1 month, and 3 months postoperatively. Clinical evaluations will include administration of a visual disturbance questionnaire (QUVID) and a satisfaction questionnaire (IOLSAT), as well as measurement of binocular and monocular visual acuities and manifest refraction.

ELIGIBILITY:
Subjects are eligible for the study if they meet the following criteria:

Note: Ocular criteria must be met in both eyes.

Inclusion Criteria:

* Undergoing uncomplicated bilateral cataract surgery with IOL implantation.
* Gender: Males and Females.
* Age: 50 years or older.
* Willing and able to provide written informed consent for participation in the study.
* Willing and able to comply with scheduled visits and other study procedures.
* Motivated for greater degree of spectacle independence vs monofocal IOL.
* Axial length ≥24.5mm in both eyes.
* Planned cataract removal by femtosecond laser.

Exclusion Criteria:

If any of the following exclusion criteria are applicable to the subject or either eye, the subject should not be enrolled in the study.

* Ocular comorbidity that might hamper postoperative visual acuity.
* Previous refractive surgery.
* Irregular corneal astigmatism.
* Evidence of keratoconus as per Pentacam.
* Expected post-op VA worse than 20/25 (Snellen).
* Refractive lens exchange.
* Difficulties comprehending written or spoken English language.
* Patients with physical or intellectual disability (e.g. Down's Syndrome, Parkinson's Disease; unable to fixate).
* Clinically significant or severe ocular surface disease that would affect study measurements based on the investigator's opinion.
* Axial length <24.5mm.
* Evidence of macular pathology as per optical coherence tomography examination.

The principal investigator reserves the right to declare a patient ineligible or non-evaluable based on medical evidence that indicates they are unsuitable for the trial.

Pregnancy has a known effect on the stability of refractions and visual acuity. As such, subjects who become pregnant during the study will not be discontinued but their data may be excluded from analyses of effectiveness.

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects ≥50 years of age presenting for cataract surgery who are appropriate candidates for intraocular lens implantation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2023-09-06 (Actual); Study Completion 2023-09-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James J Wiens, MD, Principal Investigator — Dr. James J. Wiens Medical Corporation
Locations (1):
- Image Plus Laser Eye Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Eyes
Period: Overall Study
Arm/Group | Bilateral Implantation of the Vivity IOL
Started | 20; 40 Eyes
Completed | 20; 40 Eyes
Not Completed | 0; 0 Eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: Eyes
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.7 (6.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0

OUTCOME MEASURES:

1. Primary Outcome: Binocular Uncorrected Distance Visual Acuity (logMAR)
Description: Binocular uncorrected distance visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
logMAR | -0.1 (0.06)

2. Primary Outcome: Binocular Uncorrected Intermediate Visual Acuity (logMAR)
Description: Binocular uncorrected intermediate visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
logMAR | 0.01 (0.08)

3. Primary Outcome: Binocular Uncorrected Near Visual Acuity (logMAR)
Description: Binocular uncorrected near visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
logMAR | 0.21 (0.11)

4. Secondary Outcome: Prediction Error
Description: Percentage of eyes with absolute prediction error of 0.5D or less
Time Frame: 3 months postoperatively
Measure: Count of Units; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 40
Eyes | 35

5. Secondary Outcome: Binocular Corrected Distance Visual Acuity (logMAR)
Description: Binocular corrected distance visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
logMAR | -0.14 (0.06)

6. Secondary Outcome: Binocular Distance Corrected Intermediate Visual Acuity (logMAR)
Description: Binocular distance corrected intermediate visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
logMAR | -0.02 (0.06)

7. Secondary Outcome: Binocular Distance Corrected Near Visual Acuity (logMAR)
Description: Binocular distance corrected near visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
logMAR | 0.18 (0.1)

8. Secondary Outcome: Monocular Corrected Distance Visual Acuity (logMAR)
Description: Monocular corrected distance visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 40
logMAR | -0.09 (0.05)

9. Secondary Outcome: Monocular Distance Corrected Intermediate Visual Acuity (logMAR)
Description: Monocular distance corrected intermediate visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 40
logMAR | 0.05 (0.09)

10. Secondary Outcome: Monocular Distance Corrected Near Visual Acuity (logMAR)
Description: Monocular distance corrected near visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Units Other Than Participants: Eyes
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 40
logMAR | 0.32 (0.15)

11. Secondary Outcome: Manifest Refraction Spherical Equivalent
Description: Manifest refraction spherical equivalent
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: diopter (D)
Units Other Than Participants: Eyes
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
Number analyzed (Eyes) | 40
diopter (D) | 0.25 (0.37)

12. Secondary Outcome: Questionnaire
Description: Questionnaire for visual disturbance scores (QUVID)
Time Frame: 3 months postoperatively
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
Participants
  "Bothered quite a bit" or "Bothered very much" by starbursts | 2
  "Bothered quite a bit" or "Bothered very much" by halos | 0
  "Bothered quite a bit" or "Bothered very much" by glare | 2
  "Bothered quite a bit" or "Bothered very much" by haze | 1
  "Bothered quite a bit" or "Bothered very much" by blurred vision | 0
  "Bothered quite a bit" or "Bothered very much" by double vision | 0
  "Bothered quite a bit" or "Bothered very much" by dark area | 0

13. Secondary Outcome: Percentage of Participants With Spectacle Independence
Description: The Intraocular Lens Satisfaction questionnaire (IOLSAT). Subjects were asked how often they needed to wear eyeglasses to see at distance, intermediate, and near. The percentage was calculated as (# of subjects responding "Never" or "Rarely") divided by (# of subjects) times 100. A higher percentage is a better outcome.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
Participants
  Spectacle independence distance (overall) | 19
  Spectcle independence intermediate (overall) | 18
  Spectacle independence near (overall) | 8

14. Secondary Outcome: Binocular Distance-corrected Low Contrast Distance Visual Acuity (logMAR)
Description: Binocular distance-corrected low contrast distance visual acuity (logMAR)
Time Frame: 3 months postoperatively
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Bilateral Implantation of the Vivity IOL
Number analyzed (Participants) | 20
logMAR | 0.05 (0.08)

ADVERSE EVENTS:
Time Frame: 3 months postoperatively
Arm/Group | Bilateral Implantation of the Vivity IOL
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-11): https://cdn.clinicaltrials.gov/large-docs/69/NCT05210569/Prot_SAP_000.pdf